CLINICAL TRIAL: NCT06431971
Title: Estimates of the Short-term Efficacy of Talineuren (TLN) and Placebo in Patients With Parkinson Disease: A Randomized, Placebo-controlled, Double-blinded, Parallel 2-arm, Multi-centre Pilot Trial
Brief Title: Estimates of the Short-term Efficacy of Talineuren (TLN) and Placebo in Patients With Parkinson Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InnoMedica Schweiz AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIBRA (TLN/PD/2)
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talineuren (Experimental): Participants receive standard of care PD treatment + 720 mg of Talineuren i.v. weekly for 18 infusions (18 weeks).
  Interventions: Drug: Talineuren
- Placebo (Placebo Comparator): Participants receive standard of care PD treatment + placebo (0.9% NaCl) i.v. weekly for 18 infusions (18 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talineuren — Talineuren infusion weekly
  Other Names: TLN; Liposomal GM1
  Arms: Talineuren
Drug: Placebo — Placebo infusion weekly
  Other Names: 0.9% NaCl
  Arms: Placebo

SUMMARY:
This study is double-blinded placebo controlled to estimate the short-term efficacy of Talineuren. The investigational Medicinal Product (IMP) is administrated 18 times intravenously as an add-on therapy to the standard of care Parkinson medication.

Talineuren is a liposomal formulation containing GM1 (monosialotetrahexosylganglioside) as the pharmacological active substance.

The results of this pilot study are essential for the sample size calculation of a subsequent larger phase II/III trial.

DETAILED DESCRIPTION:
The ganglioside lipid GM1 (monosialotetrahexosylganglioside) has attracted attention in scientific literature as a promising neuroprotective agent. Research suggests that GM1 ganglioside holds promise not only in the treatment of neurodegenerative disorders like Parkinson disease (PD) and Alzheimer's disease but also in promoting nerve regeneration post-injury. Furthermore, investigations into its potential to improve cognitive function and memory underscore its versatility as a therapeutic agent. Numerous clinical studies have demonstrated its therapeutic potential in treating (PD) patients.

Talineuren (TLN) represents a novel approach to harnessing the therapeutic benefits of GM1. TLN is a liposomal formulation, comprising GM1 as its pharmacologically active ingredient, which is expected to cross the blood-brain barrier more efficiently as free GM1 and therefore is able to deliver more GM1 to the brain. This innovative composition is designed to optimize the neuroprotective effects of GM1.

Study Description:

This study is designed as a double-blinded, placebo-controlled trial to evaluate the short-term efficacy of TLN in PD management. The investigational Medicinal Product (IMP), TLN, is weekly intravenously administered 18 times as an add-on therapy alongside patients' current standard-of-care PD medication. Talineuren, encapsulating GM1 within liposomes, is anticipated to facilitate enhanced delivery and bioavailability of the neuroprotective agent, GM1.

Objectives:

The primary objective is to obtain statistical estimates of change from baseline and variance for TLN and placebo and to compare these between groups for MDS-UPDRS part III score in the "off" medication state (i.e. Levodopa challenge test (LCT); motor symptoms evaluated by physician).

Secondary objectives are to obtain the change from baseline and variance of TLN and placebo and compare these between the groups for :

* MDS-UPDRS total score (part I + part II + part III "off" + part IV)
* MDS-UPDRS part I (non-motor symptoms in daily life)
* MDS-UPDRS part II (motor symptoms in daily life)
* MDS-UPDRS part III "on medication"
* MDS-UPDRS total part IV (motor complications)
* Proportion of patients meeting or exceeding the minimum clinically important difference (MCID) in motor and non-motor symptoms (MDS-UPDRS) and quality of life (PDQ-39) over time
* Quality of life (PDQ-39)
* Mental condition (MoCA)
* Parkinson medication (LEDD)

Research objectives (biomarkers):

-Assessment of literature-described biomarkers (prognostic, predictive, monitoring and/or response biomarkers) pre- and post-TLN or placebo intervention.

Through evaluation and statistical analysis, this study seeks to elucidate the therapeutic potential of TLN in addressing the multifaceted challenges of Parkinson's disease. By providing insights into treatment efficacy, medication usage, symptom management, and quality of life improvements, our findings aim to inform future advancements in PD management and enhance patient care.

The results of this pilot study are essential for the sample size calculation of a subsequent larger phase II/III trial.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature.
2. Male and female subjects, aged 30 to 85 years.
3. Confirmed PD according to British brain bank criteria.
4. Hoehn and Yahr Stage 0 - 2.5 on medication.
5. Stable dopaminergic PD treatment (including DBS) for a month at least.
6. Absence of dementia confirmed by cognitive testing (MoCA ≥24).

Exclusion Criteria:

1. Previous treatment with Talineuren (i.e. participants from NEON trial are not allowed)
2. Contraindications to the class of drugs under study, e.g., known hypersensitivity or allergy to class of drugs or the investigational products.
3. Women who are pregnant or breast feeding, or planning to become pregnant during the course of the trial or in the 12 weeks following the trial.
4. Lack of safe contraception, defined as:

   * Female participants of childbearing potential, not willing to use double method of contraception (hormonal and mechanical) for the entire study duration.

   Note: Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
   * Male participants, not using and not willing to use a medically reliable method of contraception for the entire study duration, such as condoms or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
5. Other clinically significant concomitant diseases states (e.g., renal failure, hepatic dysfunction, cardiovascular disease etc.) that is are not under stable control.
6. Known or suspected non-compliance, drug or alcohol abuse.
7. Inability to follow the procedures of the trial, e.g., due to language problems, psychological disorders etc. of the participant.
8. Participation in another trial with an investigational drug within the 30 days preceding and during the present trial.
9. Enrolment of the investigator, his/her family members, employees and other dependent persons.
10. Subject has an atypical parkinsonian syndrome or secondary parkinsonism.
11. Patients with comorbidity that may interfere with the course of the trial.
12. Patients who are not considered to be eligible to participate in clinical trial by the investigator.
13. Patients in adjustment of deep brain stimulation (DBS) parameters
14. Patients with known impaired granulopoiesis

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale score | Baseline, week 7, 11, 15, 19 and 22
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) will be used by the patient and physician to evaluate various symptoms of Parkinson disease including non-motor and motor experiences of daily living and motor complications.
  The MDS-UPDRS Scale consists of 4 parts:
  * Part 1 (Nonmotor aspects of experiences of daily living) with 13 items.
  * Part 2 (Motor aspects of experiences of daily living) with 13 items.
  * Part 3 (Motor examination) with 18 items.
  * Part 4 (Motor complications) with 6 items.
  Each item is rated with 0=normal, 1=slight, 2=mild, 3=moderate, 4=severe. The lower the score, the fewer / less severe the symptoms.

SECONDARY OUTCOMES:
Parkinson disease Quality of Life Questionnaire score | Baseline, week 19
  Parkinson disease Quality of Life Questionnaire (PDQ-39) will be completed by the patient. The proportion of patients reaching or exceeding the minimal clinical important difference (MCID) will be assessed.
  This questionnaire consists of 39 items in 8 dimensions with 0 = perfect health, 100 = worse health.
Montreal Cognitive Assessment score | baseline, week 19
  Patient's mental condition is assessed using the Montreal Cognitive Assessment (MoCA) by the physician together with the patient where the patient can reach a score of 0-30. A final total score of 26 and above is considered normal.
Change in Levodopa equivalent daily dose | Through study completion, an average of 22 weeks
  Levodopa equivalent daily dose (LEDD) in [mg] will documented at each study visit.

OTHER OUTCOMES:
Number of IMP-related adverse events | From the date of the first administration until week 22
  Incidence and severity of treatment-emergent AEs (TEAEs) from the start of the treatment until the safety visit (week 22) using CTCAE criteria (V5.0).
Proportion of feasibility parameters | Up to week 22
  Collecting of information for a subsequent larger phase II trial. The following information will be assessed:
  * Acceptance proportion: the proportion of patients willing to participate in this trial
  * Drop-out proportion & reason: the proportion of enrolled subjects who pre-maturely discontinue the trial. The reason for the discontinuation shall be recorded, if possible, so to be able to identify any potential issues in the design and procedures of the trial that can be improved for the subsequent trial.
  * Failure proportion of IMP-administration: Proportion of visits that need to be rescheduled because no vein for IMP-administration is found.
Mean values of Biomarkers | Baseline, week 19
  -To detect and assess the presence of blood-derived biomarkers selected from literature at baseline and end of intervention, and to compare the obtained values in between treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologisches Institut Konolfingen, Konolfingen, Switzerland

IPD SHARING:
Plan to Share IPD: No